CLINICAL TRIAL: NCT04357288
Title: Randomized Evaluation of Decision Support Interventions for Atrial Fibrillation
Acronym: RED-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Heart Association (Other); Patient-Centered Outcomes Research Institute (Other); Mayo Clinic (Other); Northwestern University (Other); Vanderbilt University (Other); University of Michigan (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elissa Ozanne, Associate Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB_00124127
Record Dates: First submitted 2020-04-13; First posted 2020-04-22 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Shared Decision Making
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient Decision Aid (Experimental): Participants in this arm will use the Patient Decision Aid (PDA), an online education tool about atrial fibrillation designed for patient use, prior to the encounter with their provider.
  Interventions: Other: Patient Decision Aid
- Encounter Decision Aid (Experimental): Participants in this arm will use the Encounter Decision Aid (EDA), an online educational tool about atrial fibrillation designed for patient-provider use, during the encounter with their provider.
  Interventions: Other: Encounter Decision Aid
- Patient & Encounter Decision Aids (Experimental): Participants in this arm will use both the PDA & EDA as described above.
  Interventions: Other: Patient Decision Aid; Other: Encounter Decision Aid
- Standard Care (No Intervention): Participants in this arm will receive standard care, that is they will not use either the PDA or EDA.

INTERVENTIONS:
Other: Patient Decision Aid — The Patient Decision Aid (PDA) is an interactive website designed for use by a participant without the need of their clinician present. It provides information about the atrial fibrillation diagnosis, possible treatments, the effect of this diagnosis on daily life, and how to prepare for a discussion about medications with a clinician. Participants may interact with the website by inputting their health information into the stroke risk calculator or answering questions about their values, goals, thoughts, etc. that they would like to discuss with their clinician.
  Arms: Patient & Encounter Decision Aids; Patient Decision Aid
Other: Encounter Decision Aid — The Encounter Decision Aid (EDA) is an interactive website designed for use by a participant and their clinician together. Together, the clinician and participant can go through the website together and input the participant's health information into the same stroke risk calculator also in the PDA. The EDA also provides information about the diagnosis of AF, living with this diagnosis, and possible treatments, and prompts discussion of how a participant's values affects these aspects of AF.
  Arms: Encounter Decision Aid; Patient & Encounter Decision Aids

SUMMARY:
This study will compare the effectiveness of the use of a Patient Decision Aid (PDA) and an Encounter Decision Aid (EDA) on Shared Decision Making (SDM) and health outcomes for at-risk participants with Atrial Fibrillation (AF) at 6 study sites. We hypothesize the combination of the PDA and EDA will be more effective in promoting high-quality SDM and in adoption of and adherence to anticoagulation than either tool alone.

DETAILED DESCRIPTION:
Background Information:

Atrial fibrillation (AF) is the most common cardiac arrhythmia worldwide, and it continues to grow in prevalence, afflicting an estimated 3 million Americans. While treatment of AF symptoms can be resource-intensive, another source of physical, social, and economic burden is thromboembolic stroke, the major cause of morbidity and mortality for both symptomatic and asymptomatic people with AF. People with AF must decide on a stroke prevention medication (typically, Warfarin or Oral Anti-Coagulants (OACs)).

Shared Decision Making (SD) is particularly useful when decisions, such as this, are value laden and complex. Models of SDM stress clear communication of the risks and benefits of all treatment options (including no treatment) to patients, who in turn need opportunities to share their treatment preferences, relevant values, and goals of care.

Decision aids are tools designed to support both people with AF and clinicians in SDM by 1) providing accurate, balanced information; 2) clarifying patients' values; and 3) improving SDM skills.

Two types of decision aids will be evaluated in the study: a patient-centered Patient Decision Aid (PDA) and an Encounter Decision Aid for collaborative use by the clinician and patient. The PDA is intended to help people with AF prepare for the medical visit with foundational understanding and questions. The EDA is intended to promote SDM between the clinician and person with AF.

Research Design & Methods:

Through a randomized controlled trial, our study will address whether the use of a PDA, and EDA, a combination of the 2, or usual care achieves the best SDM process and health outcomes. We will assess the comparative effectiveness of those 4 approaches in terms of their ability to affect the following outcomes: 1) SDM outcomes, including decisional conflict, knowledge, and quality of patient-clinician communication; and 2) health outcomes, including adoption rates of anticoagulation therapy, adherence to anticoagulation therapy regimen, bleeding, stroke/systemic embolism, and death. Data collection will include medical record review, survey completion, and video/audio recording of the clinician encounter.

Study sites:

Recruitment is planned to occur from 6 sites within the US.

Data Collection:

Self-reported outcomes from people with AF and clinicians will be collected at the end of each clinical encounter. In addition, clinicians will complete a survey that collects data on their demographics and practice characteristics.

Data from the medical record will be abstracted for all enrolled participants with AF to capture demographic, clinical, and medication prescription data.

ELIGIBILITY:
Patient Participants -

Inclusion Criteria:

1. Adults (18 and older)
2. Are diagnosed with Atrial Fibrillation
3. Are aware they have been diagnosed with Atrial Fibrillation
4. Participants with additional risk of thromboembolic events (CHA2DS2-VASc scores ≥ 1 in men and ≥ 2 in women)

Exclusion Criteria:

1. Participants deemed by their clinician or research personnel to be ineligible for consideration of taking or of foregoing anticoagulation
2. Have deficits in cognitive abilities or sensory input
3. Have a language barrier significant enough to impede shared decision making and/or the provision of written informed consent.

Clinician Participants -

Inclusion Criteria:

1. All clinicians (MDs, NP/PAs, PharmDs, APPs, etc.) that are responsible for the modality of Anticoagulation in eligible AF patients at participating sites, without exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1117 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | Post encounter surveys will be given or sent within 1 week after the visit
  Validated scale of 16 questions that evaluates 1) uncertainty in making a healthcare decision, 2) factors contributing to the uncertainty, and 3) the participant's perceived effective decision making. Answers range in a 5 point Likert scale from 0=strongly agree to 4=strongly disagree. Clarity and understanding are indicated if the participant "strongly agrees" to the statements, so smaller scores are better.
Patient Knowledge | Post encounter surveys will be given or sent within 1 week after the visit
  An 8-question survey assesses a participant's knowledge about atrial fibrillation and anticoagulation use after the intervention. Participants not in the intervention arm will also take this survey for comparison. Each question uses a response format of "true / false / do not know". All questions are answered with full access to the decision aid(s) (if not in standard care arm) since they are not meant to test recall. "Better" scores will be measured by how many questions that a participant answers correctly.
Shared Decision Making | Post encounter surveys will be given or sent within 1 week after the visit
  The extent of shared decision making between the participant and provider that took place during the encounter will be assessed by study team members using the Observing Patient Involvement scale (OPTION12). The scale consists of 12 items scored from 0, "the behavior is not observed," to 4, "the behavior is observed and executed to a high standard." The more shared decision making behaviors observed the better, so a higher score is "better" for this scale.

SECONDARY OUTCOMES:
Decision Regret | Survey will be given at 6 months after enrollment and again at 12 months after enrollment
  Decision Regret will be assessed by asking participants to reflect on the decision they made about taking a blood thinner and/or which blood thinner to take after their encounter with their clinician. The measure consists of 5 items assessed on a 5-point Likert scale from "Strongly agree" to "Strongly disagree".
Preparation for Decision Making | Post encounter surveys will be given or sent within 1 week after the visit
  Preparation for Decision Making Scale is a validated scale which will assess participants' perspectives of the tools' usefulness in preparing them to communicate with their clinicians and for Shared Decision Making. These questions are answered on a Likert scale ranging from 1=not at all to 5=a great deal. A higher score indicates that they are better prepared and, thus, a better outcome.
Quality of Communication | Post encounter surveys will be given or sent within 1 week after the visit
  The Quality of Communication survey is a 3-item modified version of the CAHPS Clinician and Group survey to determine the extent to which communication is patient-centered, contains technical information that is easily understood, and is respectful. Each item is assessed on a 3-point scale that will be individually reported: 1=Yes, definitely; 2=Yes, somewhat; and 3=No. The more 1's that are chosen indicates the higher quality of communication and, thus, a better outcome.
9-item Shared Decision Making Questionnaire (SDMQ9) | Post encounter surveys will be given or sent within 1 week after the visit
  The SDMQ9 assesses the quality of participant involvement in the process of decision-making with their clinician from the perspective of the participant. Each item is assessed on a 6-point Likert scale from "completely disagree" to "completely agree". Clarity and knowledge would be indicated by "completely agree", so a higher score is "better".
Control Preference Scale | Post encounter surveys will be given or sent within 1 week after the visit
  This scale assesses participants' desire to participate in Shared Decision Making. This scale is an adaptation of the Degner & Sloan's Control Preference Scale. It is a one item question that asks people if they want to make the decision alone, with their clinician, or have their clinician make it. There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Patient Satisfaction with the Decision Aid | Post encounter surveys will be given or sent within 1 week after the visit; again at 6 months; and again at 12 months
  This will be assessed with 5 questions. Participants will be asked questions about if they used the PDA before their appointment, used the PDA during their appointment, their likelihood to recommend the PDA, the amount of information presented, and if the PDA seemed biased. There is no "better" or more correct answer; it is up to the patient's opinion.
Collaborative Agreement | Post encounter surveys will be given or sent within 1 week after the visit
  Collaborative agreement will assess decision concordance between the participant and the clinician. Both the participant and clinician will be asked to report about what decision (anticoagulation no/yes-which one) was made during the index visit. Decisions will also be abstracted from Electronic Health Records and through assessment of audiovisual recordings by research staff. Agreement will be calculated between all four sources and reported. There is no "better" score besides how many answers line up between the clinician and the patient; we are measuring understanding between them.
Anticoagulation Adherence 1 - Visual Analogue Scale | Survey will be given at 6 months after enrollment and again at 12 months after enrollment
  Anticoagulation Adherence 1 will be assessed by a 100-point visual analogue scale (VAS) where participants indicate the percentage of medication taken since prior visit. This ranges from 0% (did not take any of their medication as prescribed) to 100% (took all of their medication as prescribed). A "better" score would be indicated on how close to 100%, as the patient should be taking the medication as prescribed by their clinician.
Anticoagulation Adherence 2 - Self-Report | Survey will be given at 6 months after enrollment and again at 12 months after enrollment
  A self-reported 7-day recall of pill-taking behavior. This asks participants whether they forgot to take any of their doses of medication (as prescribed). If they answer yes, they indicate the number of tablets missed per day, per week, and/or per month. Then they are asked how many pills they skipped in the past 7 days. They are asked how many days in the past week that they took more than the prescribed dosage of drug. The are asked if they had any side effects from their drugs, and if yes, what those side effects were. They are asked if they missed any doses due to the side effects. They are asked if the cost of their medication affected taking it. Finally, they are asked how taking their medication has changed their life.
Anticoagulation Adherence 3 - Warfarin Use | We gather this information throughout the length of the participant's enrollment (approximately 12 months)
  For participants who choose to stay on Warfarin, we will also use as a measure of adherence: the proportion of international normalized ration (INR) tests obtained/scheduled. This includes 2 questions: was the patient on Warfarin prior to enrollment, and were INR measures taken after enrollment.
Anticoagulation Adherence 4 - Time in Therapeutic Range | We gather this information throughout the length of the participant's enrollment (approximately 12 months)
  For participants who choose to stay on Warfarin, we will also use as a measure of adherence Time in Therapeutic Range. This is the duration of time in which the patients International Normalized Ratio (INR) is in the target range, typically values between 2 - 3. (INR is a blood test administered by the clinician to determine the patient's anticoagulation control.)
Treatment Choice | Post encounter surveys will be given or sent within 1 week after the visit; again at 6 months; and again at 12 months
  Treatment Choice will be assessed by asking participants to identify which treatment (drug) they chose and if their decisions would be different if there were no out-of-pocket costs.
Fidelity of Decision Aids | Post encounter surveys will be given or sent within 1 week after the visit
  Fidelity of SDM Tool by the clinician will be assessed by a review of the recording looking for key items to be addressed. A checklist of key elements will be assessed in all four arms to assess not only the fidelity but potential contamination. A sum of the components in the checklist will be calculated for each recording and compared across arms. There is no "better" score; we are measuring how they use the Decision Aid.
Clinical Events | Survey will be given and data will be collected at 12 months after enrollment
  Strokes and bleeds requiring medical assistance will be monitored. Because very few of these are expected, we will rely on participant/clinician self-report and medical record review 12 months post enrollment for each participant. Chart review will include identification of clinical event outcomes: death, stroke, systemic embolism, transient ischemic attack clinically-relevant non-major bleeding, and major bleeding.
Encounter Length | Post encounter surveys will be given or sent within 1 week after the visit
  Encounter Length will be assessed by comparing the length in minutes of the discussion about anticoagulation and of the office visit between the different arms, when available. Study notes and video/audio records will be used to assess encounter length.
Min/Max Scale | Post encounter surveys will be given or sent within 1 week after the visit
  1-item instrument that determines if patients have minimizer or maximizer tendencies. Medical minimizers are individuals who prefer to do as little as possible when it comes to medicine and their health, whereas medical maximizers prefer active and aggressive medical treatments and being proactive about their health. There is no "better" score; it is up to patient opinion.
Anticoagulation Persistence | Approximately 12 months after enrollment
  Anticoagulation persistence: Using data from pharmacy refills, we will calculate anticoagulation persistence throughout enrollment using the percent days covered (PDC) based on prescription refill behaviors (total days supply of anticoagulant filled / total days of observation from the first prescription fill date; range 0-100%). We will also pull all pharmacy refills for the 12 months prior to enrollment. This will allow us to calculate persistence for prior use of anticoagulants for the review cohort to compare to persistence post encounter and see if there is an impact.
Medical History | We gather medical information at the time of enrollment; again at 6 months; and again at 12 months after enrollment.
  Medical history relevant to study aims will be collected will be physiological parameters: such as hypertension, congestive heart failure, rheumatic heart disease, prior heart valve replacement, implantable cardiac device, deep vein thrombosis/pulmonary embolism, prior cerebrovascular events, diabetes mellitus, chronic renal disease, liver disease, coronary artery disease, peripheral arterial disease, prior major bleeding or predisposition to bleeding, medication usage predisposing to bleeding, alcohol use, medication prescribed during enrollment visit, concomitant medications, prior use of systematic anticoagulation for any reason, and INR measures (if the patient was on Warfarin previously, if INR measures were taken after enrollment).
Adapted Illness Intrusiveness Ratings | Post encounter surveys will be given or sent within 1 week after the visit; again at 6 months; and again at 12 months
  This will be collected using a modified version of the Illness Intrusiveness Ratings Scale, a 13-item self-report instrument. The AIIR assesses the extent to which disease and treatment interfere with meaningful daily living among people affected by chronic disease. Answers range from 1=Not very much to 7=very much. A lower score is "better" because it would indicate that their daily life is not bothered very much by their choice of treatment.
Values Trade-off | Post encounter surveys will be given or sent within 1 week after the visit
  1-item instrument that assesses patient preference of either taking a stroke prevention drug every day, which has a risk of causing serious bleeding, or not taking a stroke prevention drug every day, even though stroke risk is higher. There is no "better" answer; it is up to patient opinion.
Clinician Satisfaction | Post encounter surveys will be given or sent within 1 week after each visit
  This will be assessed with 6 questions answered by a 5-point Likert scale questioning satisfaction with discussion about anticoagulation medication choice. Answers range from 1=not at all satisfied to 5=completely satisfied. The clinician will also be asked whether they would recommend the approach used to other clinicians for other discussions on with a "yes/no/not sure" answer format. A lower score would indicate higher satisfaction, so lower is "better".
Choice of Anticoagulant | Post encounter surveys will be given or sent within 1 week after the visit; again at 6 months; and again at 12 months
  We will review the electronic medical record (EMR), patient- and clinician-reported choice, and recordings of the visit to determine the prescribed anticoagulant and whether and when switches to another agent or to no anticoagulant took place. Together, they should capture choice and switches even when these occur as a result of changes in clinician (e.g., from cardiology to primary care). When available, we will note the documented reasons from clinical notes for choosing and switching as well as with which clinician the change was made (e.g primary, cardiology, etc.).
Predicting Mortality and Healthcare Utilization (Quality of Life) | Post encounter surveys will be given or sent within 1 week after the visit; again at 6 months; and again at 12 months
  1-item instrument that assesses patient self-reported health on a scale from 1 = "poor" to 5 = "excellent", which predicts mortality, hospitalization, and high outpatient use.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Ozanne, PhD, Principal Investigator — University of Utah; Angela Fagerlin, PhD, Study Director — University of Utah
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - The Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
We will follow the funders' open-data policies.
Time Frame: We will follow the funders' open-data policies.
Access Criteria: We will follow the funders' open-data policies.
URL: https://professional.heart.org/en/research-programs/aha-research-policies-and-awardee-hub/open-science-policy-statements-for-aha-funded-research

REFERENCES:
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Elwyn G, Hutchings H, Edwards A, Rapport F, Wensing M, Cheung WY, Grol R. The OPTION scale: measuring the extent that clinicians involve patients in decision-making tasks. Health Expect. 2005 Mar;8(1):34-42. doi: 10.1111/j.1369-7625.2004.00311.x. PMID 15713169
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Background] Agency for Healthcare Research and Quality. CAHPS Clinician & Group Survey. 2018.
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Degner LF, Sloan JA. Decision making during serious illness: what role do patients really want to play? J Clin Epidemiol. 1992 Sep;45(9):941-50. doi: 10.1016/0895-4356(92)90110-9. PMID 1432023
- [Background] O'Connor A, Cranney A. User Manual - Acceptability [document on internet]. 1996.
- [Background] O'Connor AM, Cranney A. Sample Tool : Acceptability ( Osteoporosis Therapy ). https://decisionaid.ohri.ca/docs/develop/Tools/Acceptability_osteoporosis.pdf. Published 1996.
- [Background] Sevilla-Cazes J, Finkleman BS, Chen J, Brensinger CM, Epstein AE, Streiff MB, Kimmel SE. Association Between Patient-Reported Medication Adherence and Anticoagulation Control. Am J Med. 2017 Sep;130(9):1092-1098.e2. doi: 10.1016/j.amjmed.2017.03.038. Epub 2017 Apr 26. PMID 28454906
- [Background] Haynes RB, Taylor DW, Sackett DL, Gibson ES, Bernholz CD, Mukherjee J. Can simple clinical measurements detect patient noncompliance? Hypertension. 1980 Nov-Dec;2(6):757-64. doi: 10.1161/01.hyp.2.6.757. PMID 7007235
- [Background] Kaatz S, Ahmad D, Spyropoulos AC, Schulman S; Subcommittee on Control of Anticoagulation. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26. doi: 10.1111/jth.13140. No abstract available. PMID 26764429
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Kim MH, Johnston SS, Chu BC, Dalal MR, Schulman KL. Estimation of total incremental health care costs in patients with atrial fibrillation in the United States. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):313-20. doi: 10.1161/CIRCOUTCOMES.110.958165. Epub 2011 May 3. PMID 21540439
- [Background] Naccarelli GV, Varker H, Lin J, Schulman KL. Increasing prevalence of atrial fibrillation and flutter in the United States. Am J Cardiol. 2009 Dec 1;104(11):1534-9. doi: 10.1016/j.amjcard.2009.07.022. PMID 19932788
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] McGrath ER, Kapral MK, Fang J, Eikelboom JW, Conghaile Ao, Canavan M, O'Donnell MJ; Investigators of the Ontario Stroke Registry. Association of atrial fibrillation with mortality and disability after ischemic stroke. Neurology. 2013 Aug 27;81(9):825-32. doi: 10.1212/WNL.0b013e3182a2cc15. Epub 2013 Jul 31. PMID 23902702
- [Background] Wolf PA, Dawber TR, Thomas HE Jr, Kannel WB. Epidemiologic assessment of chronic atrial fibrillation and risk of stroke: the Framingham study. Neurology. 1978 Oct;28(10):973-7. doi: 10.1212/wnl.28.10.973. PMID 570666
- [Background] Conen D, Chae CU, Glynn RJ, Tedrow UB, Everett BM, Buring JE, Albert CM. Risk of death and cardiovascular events in initially healthy women with new-onset atrial fibrillation. JAMA. 2011 May 25;305(20):2080-7. doi: 10.1001/jama.2011.659. PMID 21610240
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation: a major contributor to stroke in the elderly. The Framingham Study. Arch Intern Med. 1987 Sep;147(9):1561-4. PMID 3632164
- [Background] Lin HJ, Wolf PA, Kelly-Hayes M, Beiser AS, Kase CS, Benjamin EJ, D'Agostino RB. Stroke severity in atrial fibrillation. The Framingham Study. Stroke. 1996 Oct;27(10):1760-4. doi: 10.1161/01.str.27.10.1760. PMID 8841325
- [Background] Tu HT, Campbell BC, Christensen S, Collins M, De Silva DA, Butcher KS, Parsons MW, Desmond PM, Barber PA, Levi CR, Bladin CF, Donnan GA, Davis SM; Echoplanar Imaging Thrombolytic Evaluation Trial (EPITHET) Investigators. Pathophysiological determinants of worse stroke outcome in atrial fibrillation. Cerebrovasc Dis. 2010;30(4):389-95. doi: 10.1159/000316886. Epub 2010 Aug 5. PMID 20693794
- [Background] Go AS, Hylek EM, Chang Y, Phillips KA, Henault LE, Capra AM, Jensvold NG, Selby JV, Singer DE. Anticoagulation therapy for stroke prevention in atrial fibrillation: how well do randomized trials translate into clinical practice? JAMA. 2003 Nov 26;290(20):2685-92. doi: 10.1001/jama.290.20.2685. PMID 14645310
- [Background] Hart RG, Benavente O, McBride R, Pearce LA. Antithrombotic therapy to prevent stroke in patients with atrial fibrillation: a meta-analysis. Ann Intern Med. 1999 Oct 5;131(7):492-501. doi: 10.7326/0003-4819-131-7-199910050-00003. PMID 10507957
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Background] Budnitz DS, Lovegrove MC, Shehab N, Richards CL. Emergency hospitalizations for adverse drug events in older Americans. N Engl J Med. 2011 Nov 24;365(21):2002-12. doi: 10.1056/NEJMsa1103053. PMID 22111719
- [Background] Boehringer-Ingelheim. Dabigatran prescribing information. http://docs.boehringer-ingelheim.com/Prescribing Information/PIs/Pradaxa/Pradaxa.pdf. Published 2017. Accessed January 8, 2018.
- [Background] Daichii Sankyo Inc. Edoxaban prescribing information. http://dsi.com/prescribing-information-portlet/getPIContent?productName=Savaysa&inline=true. Published 2017. Accessed January 8, 2018.
- [Background] Janssen Pharmaceuticals Inc. Rivaroxaban prescribing information. https://www.xareltohcp.com/shared/product/xarelto/prescribing-information.pdf. Published 2011. Accessed January 8, 2018.
- [Background] Bristol-Myers Squibb Company. Apixaban prescribing information. https://packageinserts.bms.com/pi/pi_eliquis.pdf. Published 2016. Accessed January 8, 2017.
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Background] Graham DJ, Reichman ME, Wernecke M, Zhang R, Southworth MR, Levenson M, Sheu TC, Mott K, Goulding MR, Houstoun M, MaCurdy TE, Worrall C, Kelman JA. Cardiovascular, bleeding, and mortality risks in elderly Medicare patients treated with dabigatran or warfarin for nonvalvular atrial fibrillation. Circulation. 2015 Jan 13;131(2):157-64. doi: 10.1161/CIRCULATIONAHA.114.012061. Epub 2014 Oct 30. PMID 25359164
- [Background] Jowett S, Bryan S, Mant J, Fletcher K, Roalfe A, Fitzmaurice D, Lip GY, Hobbs FD. Cost effectiveness of warfarin versus aspirin in patients older than 75 years with atrial fibrillation. Stroke. 2011 Jun;42(6):1717-21. doi: 10.1161/STROKEAHA.110.600767. Epub 2011 Apr 21. PMID 21512184
- [Background] Dorian P, Kongnakorn T, Phatak H, Rublee DA, Kuznik A, Lanitis T, Liu LZ, Iloeje U, Hernandez L, Lip GY. Cost-effectiveness of apixaban vs. current standard of care for stroke prevention in patients with atrial fibrillation. Eur Heart J. 2014 Jul 21;35(28):1897-906. doi: 10.1093/eurheartj/ehu006. Epub 2014 Feb 9. PMID 24513791
- [Background] Harrington AR, Armstrong EP, Nolan PE Jr, Malone DC. Cost-effectiveness of apixaban, dabigatran, rivaroxaban, and warfarin for stroke prevention in atrial fibrillation. Stroke. 2013 Jun;44(6):1676-81. doi: 10.1161/STROKEAHA.111.000402. Epub 2013 Apr 2. PMID 23549134
- [Background] Limone BL, Baker WL, Kluger J, Coleman CI. Novel anticoagulants for stroke prevention in atrial fibrillation: a systematic review of cost-effectiveness models. PLoS One. 2013 Apr 23;8(4):e62183. doi: 10.1371/journal.pone.0062183. Print 2013. PMID 23626785
- [Background] Lee S, Anglade MW, Pham D, Pisacane R, Kluger J, Coleman CI. Cost-effectiveness of rivaroxaban compared to warfarin for stroke prevention in atrial fibrillation. Am J Cardiol. 2012 Sep 15;110(6):845-51. doi: 10.1016/j.amjcard.2012.05.011. Epub 2012 May 30. PMID 22651881
- [Background] Freeman JV, Zhu RP, Owens DK, Garber AM, Hutton DW, Go AS, Wang PJ, Turakhia MP. Cost-effectiveness of dabigatran compared with warfarin for stroke prevention in atrial fibrillation. Ann Intern Med. 2011 Jan 4;154(1):1-11. doi: 10.7326/0003-4819-154-1-201101040-00289. Epub 2010 Nov 1. PMID 21041570
- [Background] Shah SV, Gage BF. Cost-effectiveness of dabigatran for stroke prophylaxis in atrial fibrillation. Circulation. 2011 Jun 7;123(22):2562-70. doi: 10.1161/CIRCULATIONAHA.110.985655. Epub 2011 May 23. PMID 21606397
- [Background] Kamel H, Johnston SC, Easton JD, Kim AS. Cost-effectiveness of dabigatran compared with warfarin for stroke prevention in patients with atrial fibrillation and prior stroke or transient ischemic attack. Stroke. 2012 Mar;43(3):881-3. doi: 10.1161/STROKEAHA.111.641027. Epub 2012 Feb 3. PMID 22308255
- [Background] Steinberg BA, Gao H, Shrader P, Pieper K, Thomas L, Camm AJ, Ezekowitz MD, Fonarow GC, Gersh BJ, Goldhaber S, Haas S, Hacke W, Kowey PR, Ansell J, Mahaffey KW, Naccarelli G, Reiffel JA, Turpie A, Verheugt F, Piccini JP, Kakkar A, Peterson ED, Fox KAA; GARFIELD-AF; ORBIT-AF Investigators. International trends in clinical characteristics and oral anticoagulation treatment for patients with atrial fibrillation: Results from the GARFIELD-AF, ORBIT-AF I, and ORBIT-AF II registries. Am Heart J. 2017 Dec;194:132-140. doi: 10.1016/j.ahj.2017.08.011. Epub 2017 Aug 24. PMID 29223431
- [Background] Ogilvie IM, Newton N, Welner SA, Cowell W, Lip GY. Underuse of oral anticoagulants in atrial fibrillation: a systematic review. Am J Med. 2010 Jul;123(7):638-645.e4. doi: 10.1016/j.amjmed.2009.11.025. PMID 20609686
- [Background] Gallagher AM, Rietbrock S, Plumb J, van Staa TP. Initiation and persistence of warfarin or aspirin in patients with chronic atrial fibrillation in general practice: do the appropriate patients receive stroke prophylaxis? J Thromb Haemost. 2008 Sep;6(9):1500-6. doi: 10.1111/j.1538-7836.2008.03059.x. Epub 2008 Jun 28. PMID 18573187
- [Background] Hylek EM, Evans-Molina C, Shea C, Henault LE, Regan S. Major hemorrhage and tolerability of warfarin in the first year of therapy among elderly patients with atrial fibrillation. Circulation. 2007 May 29;115(21):2689-96. doi: 10.1161/CIRCULATIONAHA.106.653048. Epub 2007 May 21. PMID 17515465
- [Background] Kon AA, Ackerson L, Lo B. How pediatricians counsel parents when no "best-choice" management exists: lessons to be learned from hypoplastic left heart syndrome. Arch Pediatr Adolesc Med. 2004 May;158(5):436-41. doi: 10.1001/archpedi.158.5.436. PMID 15123475
- [Background] Byrne PJ, Murphy A. Informed consent and hypoplastic left heart syndrome. Acta Paediatr. 2005 Sep;94(9):1171-5. doi: 10.1111/j.1651-2227.2005.tb02069.x. PMID 16203668
- [Background] Moyer A, Salovey P. Patient participation in treatment decision making and the psychological consequences of breast cancer surgery. Womens Health. 1998 Summer;4(2):103-16. PMID 9659000
- [Background] Haynes RB, McKibbon KA, Kanani R. Systematic review of randomised trials of interventions to assist patients to follow prescriptions for medications. Lancet. 1996 Aug 10;348(9024):383-6. doi: 10.1016/s0140-6736(96)01073-2. PMID 8709739
- [Background] Street RL Jr, Voigt B. Patient participation in deciding breast cancer treatment and subsequent quality of life. Med Decis Making. 1997 Jul-Sep;17(3):298-306. doi: 10.1177/0272989X9701700306. PMID 9219190
- [Background] Krug S. Rocket Surgery Made Easy: The Do-It Yourself Guide to Finding and Fixing Usability Problems. Berkley, CA: New Riders; 2010.
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Siouta E, Hellstrom Muhli U, Hedberg B, Brostrom A, Fossum B, Karlgren K. Patients' experiences of communication and involvement in decision-making about atrial fibrillation treatment in consultations with nurses and physicians. Scand J Caring Sci. 2016 Sep;30(3):535-46. doi: 10.1111/scs.12276. Epub 2015 Dec 28. PMID 26709843
- [Background] Mann DM, Ponieman D, Montori VM, Arciniega J, McGinn T. The Statin Choice decision aid in primary care: a randomized trial. Patient Educ Couns. 2010 Jul;80(1):138-40. doi: 10.1016/j.pec.2009.10.008. Epub 2009 Dec 2. PMID 19959322
- [Background] Montori VM, Shah ND, Pencille LJ, Branda ME, Van Houten HK, Swiglo BA, Kesman RL, Tulledge-Scheitel SM, Jaeger TM, Johnson RE, Bartel GA, Melton LJ 3rd, Wermers RA. Use of a decision aid to improve treatment decisions in osteoporosis: the osteoporosis choice randomized trial. Am J Med. 2011 Jun;124(6):549-56. doi: 10.1016/j.amjmed.2011.01.013. PMID 21605732
- [Background] Weymiller AJ, Montori VM, Jones LA, Gafni A, Guyatt GH, Bryant SC, Christianson TJ, Mullan RJ, Smith SA. Helping patients with type 2 diabetes mellitus make treatment decisions: statin choice randomized trial. Arch Intern Med. 2007 May 28;167(10):1076-82. doi: 10.1001/archinte.167.10.1076. PMID 17533211
- [Background] Mullan RJ, Montori VM, Shah ND, Christianson TJ, Bryant SC, Guyatt GH, Perestelo-Perez LI, Stroebel RJ, Yawn BP, Yapuncich V, Breslin MA, Pencille L, Smith SA. The diabetes mellitus medication choice decision aid: a randomized trial. Arch Intern Med. 2009 Sep 28;169(17):1560-8. doi: 10.1001/archinternmed.2009.293. PMID 19786674
- [Derived] Ozanne EM, Barnes GD, Brito JP, Cameron KA, Cavanaugh KL, Greene T, Jackson EA, Montori VM, Steinberg BA, Witt DM, Noseworthy P, Passman RS, Kansal P, Crossley G, Roden DM, Christensen JT, Ariotti A, Jones AE, Bardsley T, Wu C, Fagerlin A; STEP-UP Writing Group. Effectiveness of shared decision making strategies for stroke prevention among patients with atrial fibrillation: cluster randomized controlled trial. BMJ. 2025 Jan 9;388:e079976. doi: 10.1136/bmj-2024-079976. PMID 39788611